CLINICAL TRIAL: NCT03482609
Title: The Effect of Postoperative Referred Pain in the Left Shoulder on Short-term Outcomes for Laparoscopic Gastrectomy- A Prospective Cohort Study
Brief Title: The Effect of Postoperative Referred Pain in the Left Shoulder on Short-term Outcomes for Laparoscopic Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Other Study IDs: FujianMU
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to explore the effect of postoperative referred pain in the left shoulder on short-term outcomes for laparoscopic gastrectomy

DETAILED DESCRIPTION:
A prospective cohort study will be performed to explore the effect of postoperative referred pain in the left shoulder on short-term outcomes for laparoscopic（including robot assisted laparoscopic surgery） gastrectomy .The evaluation parameters are overall postoperative morbidity rates,perioperative clinical efficacy and 3-year survival and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years
* Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* cT1-4a, N0-3, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
* No distant metastasis is observed. And the spleen, pancreas or other adjacent organs are not involved by the tumor.
* Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
* American Society of Anesthesiology score (ASA) class I, II, or III
* Written informed consent

Exclusion Criteria:

* patients whose previous history of chronic shoulder pain
* Women during pregnancy or breast-feeding
* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* Enlarged or bulky regional lymph node envelop important vessels
* History of other malignant disease within past five years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* History of continuous systematic administration of corticosteroids within one month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of predicted values
* Difficulty of understanding V A S(Visual Analogues Score).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergoing laparoscopic (including robot assisted laparoscopic surgery) radical gastrectomy for gastric cancer are included.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative referred pain in the left shoulder within 1 month | 30 days
  The incidence of postoperative referred pain in the left shoulder within 1 month

SECONDARY OUTCOMES:
overall postoperative morbidity rates | 30 days
  overall postoperative morbidity rates
3-year disease overall survival rate | 36 months
  3-year disease overall survival rate
3-year disease free survival rate | 36 months
  3-year disease free survival rate
3-year recurrence pattern | 36 months
  3-year recurrence pattern
intraoperative morbidity rates | 1 day
  The intraoperative morbidity rates are defined as the rates of event observed within operation.
overall postoperative serious morbidity rates | 30 days
  overall postoperative serious morbidity rates
postoperative recovery course | 30 days
  postoperative recovery course
postoperative nutritional status and quality of life | 30 days
  postoperative nutritional status and quality of life
inflammatory and immune response | 7 days
  inflammatory and immune response

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, professor, Principal Investigator — Fujian Medical University Union Hospital,China
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No